CLINICAL TRIAL: NCT02348242
Title: Ocular Surface Disorders in Patients in Intensive Care Units, a Comparative Study
Brief Title: Ocular Surface Disorders in Patients in Intensive Care Units, a Comparative Study of Three Preventive Approaches
Acronym: OCUREA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-A01197-40
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Corneal Diseases
Keywords: Intensive care; corneal damage; prevention; nursing protocol
MeSH Terms: conditions — Corneal Diseases; Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aqueous gel (Experimental): In the same patient : one eye receives regular administration of aqueous gel (experimental treatment 1) and the other eye receives regular administration of artificial tears (active comparator)
  Interventions: Device: Aqueous Gel; Device: Artificial Tears
- Eyelid occlusion dressing (Experimental): In the same patient : one eye is closed with an eyelid closure dressing (experimental treatment 2) and the other eye receives regular administration of artificial tears (active comparator)
  Interventions: Device: Eyelid Occlusion Dressing; Device: Artificial Tears

INTERVENTIONS:
Device: Aqueous Gel — 1 drop of Dexpanthenol® 0.2% aqueous gel in the eye every 6 hours
  Other Names: Dexpanthenol® 0.2%
  Arms: Aqueous gel
Device: Eyelid Occlusion Dressing — Eyelid occlusion using pro-ophta® eyelid occlusion dressing, dressing to be verified every 6 hours and replaced daily
  Other Names: Pro-Ophta® Dressing
  Arms: Eyelid occlusion dressing
Device: Artificial Tears — 1 drop of Phylarm® artificial tears in the eye every 6 hours
  Other Names: Phylarm®

SUMMARY:
60% of the patients hospitalized in intensive care and sedated suffer from insufficient inferior eyelid occlusion. Thus, they are at risk for corneal damage (estimated risk 20% to 57%). The prevention of such corneal damage can be done using several techniques (artificial tears, eyelid occlusion dressing, aqueous gel). The efficacy of these techniques has never been compared in a rigorous study. Therefore it is not yet possible to determine an evidence-based strategy to prevent corneal damage in intensive care patients.

This study aims at assessing the efficacy of primary prevention of corneal lesions in intensive care patients, in order to elaborate an evidence-based nursing protocol.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* hospitalized in an intensive care unit
* tracheal intubation and mechanical ventilation since less than 24 hours, with an expected duration of artificial ventilation superior to 72h

Exclusion Criteria:

* Patient currently treated by eyedrops for glaucoma
* antecedent of corneal transplant
* ocular prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Incidence rate of corneal lesions (grade > 0 in the Mercieca classification) | participants will be followed for the duration of stay in intensive care unit, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel DEVYS, Dr, Principal Investigator — Fondation Ophtalomologique Adolphe de Rothschild
Locations (1):
- Fondation ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France